CLINICAL TRIAL: NCT01031680
Title: A 24-week, Multicentre, Randomised, Double-blind, Age-stratified, Placebo Controlled, Phase III Study With a 80-week Extension Period to Evaluate the Efficacy and Safety of Dapagliflozin 10 mg Once Daily in Pts With T2DM, CV Disease and Hypertension Who Exhibit Inadequate Glycaemic Control on Usual Care
Brief Title: Efficacy and Safety in Patients With Type 2 Diabetes Mellitus, Cardiovascular Disease and Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1690C00018
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Disease; Hypertension; Inadequate Glycaemic Control
Keywords: dapagliflozin; diabetes; cardiovascular disease; hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Hypertension; Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Dapagliflozin 10 mg tablet
  Interventions: Drug: Dapagliflozin
- 2 (Placebo Comparator): Matching placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg tablet, oral, once daily, 24- week treatment and 80-week extension period
  Arms: 1
Drug: Placebo — Matching placebo tablet, oral, once daily, 24- week treatment and 80-week extension period
  Arms: 2

SUMMARY:
This study is carried out to assess whether dapagliflozin lowers blood glucose, body weight and blood pressure, when added to patients existing medications and how it compares with their usual treatment without added dapagliflozin. Safety data will be collected and analysed to confirm that treatment with dapagliflozin is safe and well tolerated in patients who have diabetes, cardiovascular disease and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus.
* Cardiovascular disease
* Hypertension

Exclusion Criteria:

* Patients with type 1 diabetes or diabetes insipidus
* Patients with 3 or more oral anti-hyperglycaemic drugs with or without insulin and/or poorly controlled diabetes
* Any clinically significant illness, which would compromise the patient's safety and their participation in the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 922 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. William Cefalu, Principal Investigator — Pennington Biomedical Research Center
Locations (140):
- United States (60):
  - Research Site, Gulf Shores, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Burbank, California
  - Research Site, Garden Grove, California
  - Research Site, Huntington Park, California
  - Research Site, Lancaster, California
  - Research Site, Salinas, California
  - Research Site, San Marino, California
  - Research Site, San Ramon, California
  - Research Site, Tustin, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Waterbury, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Deerfield Beach, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Stone Mountain, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Research Site, West Monroe, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Brick, New Jersey
  - Research Site, Oradell, New Jersey
  - Research Site, New Hyde Park, New York
  - Research Site, The Bronx, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Phoenixville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Reading, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Kingsport, Tennessee
  - Research Site, Carrollton, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tomball, Texas
  - Research Site, Ogden, Utah
  - Research Site, Danville, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
- Argentina (8):
  - Research Site, La Plata, Buenos Aires
  - Research Site, Buenos Aires, Buenos Aires F.D.
  - Research Site, Caba, Buenos Aires F.D.
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Mendoza, Mendoza Province
  - Research Site, Santa Fe, Santa Fe Province
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aires
- Canada (17):
  - Research Site, Calgary, Alberta
  - Research Site, New Westminster, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Carbonear, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Courtice, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Smiths Falls, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Lachine, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Marc-des-Carrieres, Quebec
  - Research Site, Sherbrooke, Quebec
- Germany (13):
  - Research Site, Potsdam, BR
  - Research Site, Bad Nauheim
  - Research Site, Berlin
  - Research Site, Erdmannhausen
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Heilbronn
  - Research Site, Hildesheim
  - Research Site, Mainz
  - Research Site, Münster
  - Research Site, Potsdam
  - Research Site, Speyer
  - Research Site, Wahlstedt
- Romania (7):
  - Research Site, Brasov, Brașov County
  - Research Site, Suceava, Suceava
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Constanța
  - Research Site, Iași
  - Research Site, Sibiu
- Slovakia (14):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Dolný Kubín
  - Research Site, Komárno
  - Research Site, Košice
  - Research Site, Kysucké Nové Mesto
  - Research Site, Liptovský Hrádok
  - Research Site, Lučenec
  - Research Site, Nitra
  - Research Site, Považská Bystrica
  - Research Site, Prievidza
  - Research Site, Rimavská Sobota
  - Research Site, Ružomberok
  - Research Site, Žilina
- Spain (13):
  - Research Site, Córdoba, Andalusia
  - Research Site, Granada, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Barcelona, Catalonia
  - Research Site, Lleida, Catalonia
  - Research Site, Olot (girona), Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Majadahonda, Madrid
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, San Juan (alicante), Valencia
  - Research Site, Valencia, Valencia
- Taiwan (6):
  - Research Site, Tainan County, Taiwan
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Vietnam (2):
  - Research Site, Hanoi, Vietnam
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Cefalu WT, Leiter LA, de Bruin TW, Gause-Nilsson I, Sugg J, Parikh SJ. Dapagliflozin's Effects on Glycemia and Cardiovascular Risk Factors in High-Risk Patients With Type 2 Diabetes: A 24-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study With a 28-Week Extension. Diabetes Care. 2015 Jul;38(7):1218-27. doi: 10.2337/dc14-0315. Epub 2015 Apr 7. PMID 25852208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 10 Feb 2010, last participant for last visit for the 24-week period: 26 May 2011. This study was conducted in 4 European countries, 2 countries in Asia/the Pacific Region, The United States, Canada, and Argentina. In total 1429 participants were enrolled and 922 participants were randomized.
Pre-assignment Details: During a placebo lead-in period, participants were counselled on dietary and life-style modifications.
Groups:
- Experimental: Dapagliflozin, 10 mg tablet, oral, once daily
- Placebo Comparator: Placebo, Matching placebo tablet, oral, once daily
Period: Overall Study
Arm/Group | Experimental | Placebo Comparator
Started | 460 (Of the 460 randomized participants only 455 were included in the full analysis set.) | 462 (Of the 462 randomized participants only 459 were included in the full analysis set.)
Completed | 403 | 404
Not Completed | 57 | 58
Not completed — Adverse Event | 8 | 3
Not completed — Lost to Follow-up | 2 | 10
Not completed — Withdrawal by Subject | 12 | 16
Not completed — Death | 2 | 1
Not completed — Subject No Longer Meets Study Criteria | 26 | 17
Not completed — Poor/Non-compliance | 5 | 6
Not completed — Safety | 1 | 0
Not completed — Incorrect Enrolment | 1 | 2
Not completed — Administrative Reason by Sponsor | 0 | 1
Not completed — Various | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set defined as all randomized participants (as randomized) who received at least one dose of double-blind study medication, who have a non-missing baseline value and at least one post-baseline efficacy value for at least one efficacy variable during double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo Comparator | Total
Number analyzed (Participants) | 455 | 459 | 914
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (6.97) | 63.0 (7.66) | 62.9 (7.32)
Age, Customized [Number; unit: Participants]
  <55 | 58 | 74 | 132
  >=55 and <65 | 205 | 189 | 394
  >=65 and <75 | 164 | 165 | 329
  >=75 | 28 | 31 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 144 | 290
  Male | 309 | 315 | 624
Haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 8.18 (0.841) | 8.08 (0.802) | 8.13 (0.823)
Seated Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 133.5 (13.48) | 133.0 (13.81) | 133.2 (13.64)
Total Body Weight [Mean (Standard Deviation); unit: kg] | 92.63 (20.504) | 93.59 (19.467) | 93.11 (19.985)
Body Mass Index (BMI) [Number; unit: Participants]
  < 25 kg/m² | 29 | 30 | 59
  >= 25 kg/m² | 426 | 429 | 855
  >= 27 kg/m² | 388 | 397 | 785
  >= 30 kg/m² | 291 | 304 | 595

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c Levels
Description: To compare the glycemic efficacy of dapagliflozin 10 mg versus placebo when added to usual care in type 2 diabetes patients with cardiovascular disease and hypertension, measured as the mean change in HbA1c from baseline to week 24.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 448 | 451
Percent | -0.38 [-0.46 to -0.30] | 0.08 [0.01 to 0.16]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significant at alpha=0.025 (2-sided). A hierarchical closed testing procedure was used to control Type I error across the primary & key secondary objectives; with treatment group and stratum as effects and baseline value as covariate for each endpoint; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.56 to -0.37], Standard Error of Mean 0.0473 — with stratum = age-by-insulin use-by-time from most recent qualifying CV event

2. Primary Outcome: Proportion of Responders Meeting All Criteria of a 3-item Endpoint of Clinical Benefit
Description: To compare the clinical benefit of dapagliflozin 10 mg versus placebo when added to usual care in type 2 diabetes patients with cardiovascular disease and hypertension at week 24, measured as the proportion of responders for a 3-item endpoint of clinical benefit, defined as an absolute drop of 0.5% or more from baseline HbA1c, and a relative drop of 3% or more from baseline for total body weight, and an absolute drop of 3 mmHg or more from baseline in seated systolic blood pressure.
Time Frame: Baseline to week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 444 | 451
Percentage of participants | 11.7 [8.7 to 14.7] | 0.9 [0.0 to 1.8]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; H0: proportion(treat) minus proportion(placebo) = 0 versus the alternative HA: proportion(treat) minus proportion(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; with age-by-insulin use-by-time from most recent qualifying CV event as stratum; Risk Difference (RD) = 9.9, 95% CI 2-sided [7.0 to 12.9]

3. Secondary Outcome: Adjusted Mean Change in Seated Systolic Blood Pressure (SBP)
Description: To compare the mean change in seated systolic blood pressure from baseline to week 8 between dapagliflozin 10 mg versus placebo.
Time Frame: Baseline to Week 8
Population: Full Analysis Set, participants with non-missing baseline and Week 8 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 451 | 459
mmHg | -2.96 [-4.29 to -1.64] | -0.99 [-2.29 to 0.32]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.0126, ANCOVA — Significant at alpha=0.05 (2-sided). Primary and key secondary endpoints are tested following a hierarchical closed testing procedure; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -1.97, 95% CI 2-sided [-3.52 to -0.42], Standard Error of Mean 0.7898 — with stratum = age-by-insulin use-by-time from most recent qualifying CV event

4. Secondary Outcome: Adjusted Mean Percent Change in Body Weight
Description: To compare the mean percent change in body weight from baseline to week 24 between dapagliflozin 10 mg versus placebo.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Body Weight
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 455 | 459
Percentage of Body Weight | -2.56 [-2.88 to -2.24] | -0.30 [-0.62 to 0.03]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -2.27, 95% CI [-2.64 to -1.89], Standard Error of Mean 0.1910 — with stratum = age-by-insulin use-by-time from most recent qualifying CV event

5. Secondary Outcome: Adjusted Mean Change in Seated Systolic Blood Pressure (SBP) at Week 24 (LOCF)
Description: To compare the mean change in seated systolic blood pressure from baseline to week 24 between dapagliflozin 10 mg versus placebo.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 451 | 459
mmHg | -2.99 [-4.36 to -1.61] | -1.03 [-2.39 to 0.32]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.0174, ANCOVA — Significant at alpha=0.05 (2-sided). Key secondary endpoints are tested following a hierarchical closed testing procedure; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -1.95, 95% CI 2-sided [-3.56 to -0.34], Standard Error of Mean 0.8203 — with stratum = age-by-insulin use-by-time from most recent qualifying CV event

6. Secondary Outcome: Proportion of Participants With a Reduction From Baseline of 5% or More in Body Weight in Participants With Baseline BMI ≥27 kg/m²
Description: To compare the proportion of participants with BMI baseline ≥27 kg/m2 with a reduction from baseline of 5% or more in body weight with dapagliflozin 10 mg versus placebo from baseline to week 24. Least Squares Mean represents the percent of participants adjusted for baseline body weight and age stratum.
Time Frame: Baseline to Week 24
Population: Full analysis set; participants with baseline BMI ≥27 kg/m² and Week 24 (LOCF) body weight value
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 388 | 397
Percentage of participants | 16.5 [12.8 to 20.2] | 4.0 [2.1 to 5.9]
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Based on methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, with adjustment for baseline value and stratum (gender); Risk Difference (RD) = 12.5, 95% CI 2-sided [8.3 to 16.6], Standard Error of Mean 2.126

ADVERSE EVENTS:
Time Frame: Non-serious / serious adverse events on or after the first day and on or prior to the last day of the 24-week double-blind treatment plus 4/30 days or up to follow-up visit if earlier, or up to and including the start date of extension period if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Experimental | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 27/460 | 26/462
Other Adverse Events (participants affected / at risk) | 89/460 | 84/462
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=460) | Placebo Comparator (N=462)
Gastroenteritis (Infections and infestations) | 2 | 1
Anal Abscess (Infections and infestations) | 1 | 0
Diarrhoea Infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 1
Localised Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Septic Shock (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Abscess Limb (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 3
Cardiogenic Shock (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Diabetic Foot (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Chest Pain (General disorders) | 1 | 2
Sudden Death (General disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Ischaemic Stroke (Nervous system disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0
Arteriosclerosis Obliterans (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Vascular Occlusion (Vascular disorders) | 0 | 1
Unassigned (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=460) | Placebo Comparator (N=462)
Hypoglycemia (Endocrine disorders) | 89 | 84

LIMITATIONS AND CAVEATS:
For participants who did not complete 8 and/or 24 weeks, respectively, LOCF was used. For HbA1c: excluding data after glycemic rescue, Weight: including data after rescue, SBP: excluding data after anti-hypertensive rescue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.